CLINICAL TRIAL: NCT00497445
Title: Additional Exercise Therapy in Patients With Peripheral Arterial Disease: The Value of Supervised Exercise Therapy After Invasive Treatment of Peripheral Arterial Disease.
Brief Title: The Value of Supervised Exercise Therapy After Invasive Treatment of Peripheral Arterial Disease
Acronym: NETP-extra
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atrium Medical Center (Other)
Responsible Party: Dr. JAW Teijink, Atrium medical centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-P-62
Record Dates: First submitted 2007-07-05; First posted 2007-07-06 (Estimated); Last update posted 2009-11-06 (Estimated); Status verified 2009-11

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral arterial disease; Exercise therapy; Angioplasty; Bypass surgery
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Angioplasty; Surgical Procedures, Operative; Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Angioplasty / surgery and exercise therapy (Experimental): Angioplasty / surgery followed by supervised exercise therapy
  Interventions: Procedure: Angioplasty / surgery and exercise therapy
- Angioplasty / surgery (No Intervention): Angioplasty / surgery alone
  Interventions: Procedure: angioplasty / surgery

INTERVENTIONS:
Procedure: angioplasty / surgery — Percutaneous vascular intervention or surgery for peripheral arterial disease
  Arms: Angioplasty / surgery
Procedure: Angioplasty / surgery and exercise therapy — Percutaneous vascular intervention or surgery for peripheral arterial disease followed by supervised exercise therapy
  Arms: Angioplasty / surgery and exercise therapy

SUMMARY:
The objective of this study is to investigate what the value is of SET after a radiological or surgical intervention for peripheral arterial disease in the aorto-iliacal, femoro-popliteal and crural segments in comparison with a control group.

DETAILED DESCRIPTION:
Treatment of peripheral arterial disease consists of vascular risk factor management and, dependent on the severity of the disease, exercise therapy, and either radiological or surgical intervention. After invasive treatment, many patients keep complaints, or complaints return, despite the fact that the treated segment is still patent.

Supervised exercise therapy (SET) has been proved to be an effective treatment for patients with intermittent claudication, with a significant increase in maximal walking distance. Further, exercise therapy contributes to an improvement in quality of life, a delay in disease progression and an improvement of the vascular risk profile.

Research on SET after an invasive intervention is rare. In one study, the effect of SET after surgical treatment on walking distance was determined. The initial claudication distance increased significantly in the exercise group, compared with surgical treatment alone.

In June 2004, the Network for Exercise Therapy Parkstad (NETP) was implemented in Heerlen and its environs. The physiotherapists of this network provide community based SET according to the protocol of the Royal Dutch Society of Physiotherapy. The web based database, which is a part of the NETP, was retrospectively searched for patients who started SET within 2 months after a radiological or surgical intervention. Seventeen patients fulfilled these criteria, and after 1, 3, 6 and 12 months, there was a significant increase in both initial claudication distance (ICD) and absolute claudication distance (ACD).

The expectation is that SET, immediately offered after an invasive intervention for peripheral arterial disease, influences walking distance and quality of life. Further, a positive influence on vascular risk factors and the frequency of re-interventions is expected.

ELIGIBILITY:
Inclusion Criteria:

* PAD stage 2 or 3 according to Fontaine,
* Surgical or radiological intervention indicated

Exclusion Criteria:

* No insurance for physiotherapy,
* Insufficient command of the Dutch language,
* Serious cardiopulmonary limitations (NYHA 3-4,)
* Major amputation,
* Serious co-morbidity prohibiting physical training

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2005-12; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
maximum walking distance | one year

SECONDARY OUTCOMES:
quality of life fontaine stage ankle brachial index vascular risk factors re-interventions patency mortality. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Joep A. Teijink, PhD, MD, Principal Investigator — Atrium medical center Parkstad
Locations (1):
- Atrium Medical Center, Heerlen, PO Box 4446, Netherlands

REFERENCES:
- [Derived] Kruidenier LM, Nicolai SP, Rouwet EV, Peters RJ, Prins MH, Teijink JA. Additional supervised exercise therapy after a percutaneous vascular intervention for peripheral arterial disease: a randomized clinical trial. J Vasc Interv Radiol. 2011 Jul;22(7):961-8. doi: 10.1016/j.jvir.2011.02.017. Epub 2011 May 14. PMID 21571547